CLINICAL TRIAL: NCT04628546
Title: Pediatric Motivational mHealth Parent Training for Child Disruptive Behaviors: Pilot Randomized Clinical Trial
Brief Title: The Parenting Young Children Check-up Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Lucy (Kathleen) McGoron, Ph.D., Assistant Professor (Research), Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K01MH110600B; K01MH110600 (NIH)
Record Dates: First submitted 2020-09-28; First posted 2020-11-13 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Disruptive Behavior; Parenting
Keywords: Parenting Interventions; Parent Training; Preschool-aged Children; Technology-based intervention; Brief Intervention; Disruptive Behavior Problems
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Intervention Model Description: Twenty parents that will be randomly assigned to the intervention group (random assignment determined through a random number generator). Twenty parents will be assigned to a control condition.
Who Masked: Participant
Masking Description: Participants are randomly assigned to intervention or control and not informed which condition to which they were assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: The Parenting Young Children Check-up Initial Check-up and Text Messages; Behavioral: The Parenting Young Children Check-up Flier and Text Messages
- Assessment Only (No Intervention)

INTERVENTIONS:
Behavioral: The Parenting Young Children Check-up Initial Check-up and Text Messages — Parents assigned to the intervention condition will go through the Initial Check-up, which is a brief intervention that uses motivational content to promote use of the Parenting Young Children Check-up parenting education website. They will also receive text messages and a brochure to connect them to the parenting education website.
  Arms: Intervention
Behavioral: The Parenting Young Children Check-up Flier and Text Messages — Parents assigned to the control condition will not go through the Parenting Young Children Check-up Initial Check-up. They will only go through assessment and then see a brief flier about the Parenting Young Children. Like the intervention condition, they will also receive text messages and a brochure to connect them to the Parenting Young Children Check-up parenting education website.
  Arms: Intervention

SUMMARY:
The PYCC is a system for parents of young children (2-5 years old) with Disruptive Behavior Problems (DBPs). The program is designed with the intentions of being used a pediatric primary care visit. Parents that report elevated child behavior problems go through a three part program. First, they go through a brief intervention on a tablet (i.e., the initial check-up) to receive feedback and learn about the PYCC; the aim is to build motivation to make parenting changes and engage in the parenting young children check-up. Next, parents receive text messages to connect them to further parent training content. Finally, parent training content is delivered via a web-based resource (i.e., the PYCC website), which includes videos to teach parenting skills. In this pilot RCT, the investigators will focus on examining the impact of the brief intervention (i.e., the initial check-up). Secondarily, the investigators will examine overall impact of the whole PYCC program and use of the parenting training website.

Parents will learn about the research opportunity through select community-based organizations in Detroit, Michigan, local posting, and a local participant registry. Through a phone call, parents will complete a demographics questionnaire and the DBP screener. The investigators aim to screen 200 parents in order to enroll 40 parents in the clinical trial.

If parents report elevated DBPs and do not meet any exclusion criteria, then they will be eligible to further participate. Parents that are eligible will complete a consent form (i.e., an online information sheet) and then be randomly assigned to intervention (n = 20) or control (n = 20). Both groups will complete a brief baseline. Both groups will also learn about the Parenting Young Children Check-up (PYCC). However, the way in which they learn about the program will differ. The control group will see a brief description about the program (i.e., an online flier) and will receive a brochure for the program through the mail. The intervention group will go through the full PYCC initial check-up and also receive a brochure through the mail. Both groups will receive text messages prompting them to engage in the PYCC.

After initial participation, parents will be free to use, or not use, the Parenting Young Children Check-up web-based resource as much as they want. Parents will enter their phone number and first name when accessing the web-based content in order for use to track their engagement. All use of the web-based resource will start with "Session 1. In this, they will choose what parenting skills they want to learn. If parents go through session 1, they will be further connected to PYCC content through tailored text messages. Texts contain links to all PYCC web-based content. Parents will be able to learn content related to "Special Time," "Labeled Praise," "Family Rules," "Effective Commands," "Offering Choices," "Routines," "Removing Attention," "Logical Consequences," and "Time out." All content of the PYCC is based on evidence-based parent training program content.

The purpose of this project is evaluate the Parenting Young Children Check-up. In particular, the investigators are interested in if the initial check-up leads parents to engage in the PYCC (i.e., completing session 1 and using the parent training content on the PYCC website).

Hypotheses include:

Primary Hypothesis: The intervention group (i.e. those randomized to complete the full initial check-up) will visit the parent training website more than the control group. The investigators hypothesize that, compared to the control group, more parents in the control group with complete "session 1," and use the PYCC web-based content to learn parenting skills (i.e., more parents will use any of this content and parents will use it more frequently).

Secondary Hypothesis (a): Participants assigned to the intervention group, as compared to those in the control group, will have higher scores for all domains consistent with the Theory of Planned Behavior at follow-up.

Secondary Hypothesis (b). Participants in the intervention group will report high levels of satisfaction (i.e., >=4 on a 5-point scale).

The investigators will also explore the impact of the PYCC on reported parenting and child behavior problems. Furthermore, the investigators will explore the impact of the initial check-up on intentions to use the parent training website.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* English speaking
* Parent to a child ages 2-5
* Report their child has elevated disruptive behavior problems on the Eyberg Child Behavior Inventory
* Have Smartphone and CIAS program works on their phone

Exclusion Criteria:

* Parent report that their child has an Autism Spectrum Disorder diagnosis
* Parent report that their child has an intellectual disability
* Parent report that their child is receiving treatment of Oppositional Defiant Disorder or ADHD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Initial use of the parenting training website session 1 | 1 month
  After learning about the program, the first point of program use is session 1 (i.e., selecting parenting skill to learn first); the investigators will track if parents completed session 1 (1) or did not (0)
Use of parent training content on the PYCC website (binary; yes or no) | 1 month
  The investigators will measure if parents use the parent training content on the Parenting Young Children Check-up Website (binary; yes or no)
Number of uses of parent training content on the PYCC website | 1 month
  The investigators will track how many of the parent training content modules parents use; there are 9 different areas of training content with two modules each, thus there is a possible range of 0-18
Use of parent training content on the PYCC website (binary; yes or no) | 3 months
  The investigators will measure if parents use the parent training content on the Parenting Young
Number of uses of parent training content on the PYCC website | 3 months
  The investigators will track how many of the parent training content modules parents use; there are 9 different areas of training content with two modules each, thus there is a possible range of 0-18

SECONDARY OUTCOMES:
Change in Attitudes, norms, and perceived behavioral control; consistent with the Theory of Planned Behavior | Baseline; 1 month
  Nine items total with 3 items each taping into each of the three elements of TPB (perceived norms, attitude, behavioral control); Rated on a 5 point scale (0 = Strongly Disagree, 1 = Disagree, 2 = neither disagree nor agree, 3 = Agree, 4 =Strongly Agree)
Change in Attitudes, norms, and perceived behavioral control; consistent with the Theory of Planned Behavior | Baseline; 3 months
  Nine items total with 3 items each taping into each of the three elements of TPB (perceived norms, attitude, behavioral control); Rated on a 5 point scale (0 = Strongly Disagree, 1 = Disagree, 2 = neither disagree nor agree, 3 = Agree, 4 =Strongly Agree)
Technology Acceptance with initial check-up | Baseline;
  6 Items specific to the initial check-up derived from the technology acceptance model tapping including ease of use, usefulness, and satisfaction, 5-point scale (0 = Strongly Disagree, 1 = Disagree, 2 = neither disagree nor agree, 3 = Agree, 4 =Strongly Agree)
Technology Acceptance Parenting Young Children Check-up | 1 month
  18 Items focused on all the elements the PYCC program that are derived from the 1technology acceptance model and tap into ease of use, usefulness, and satisfaction; 5-point scale (0 = Strongly Disagree, 1 = Disagree, 2 = neither disagree nor agree, 3 = Agree, 4 =Strongly Agree)

OTHER OUTCOMES:
Change in Child Disruptive Behavior Intensity | Baseline; 1 month; 3 month
  Eyberg child behavior inventory; 36 items rated on a 7 point scale ((Never=1; Seldom=2-3; Sometimes=4; Often=5-6; Always=7))
Change in Child Disruptive Behavior Intensity | Baseline; 3 month
  Eyberg child behavior inventory; 36 items rated on a 7 point scale ((Never=1; Seldom=2-3; Sometimes=4; Often=5-6; Always=7))
Change in Child Disruptive Behavior Problems Count | Baseline; 1 month
  Eyberg child behavior inventory; 36 items rated as a problem or not (0 =no, 1 = yes)
Change in Child Disruptive Behavior Problems Count | Baseline; 3 months
  Eyberg child behavior inventory; 36 items rated as a problem or not (0 =no, 1 = yes)
Change in Parenting | Baseline; 1 months
  The Alabama Parenting Questionnaire; 31 items rated on a 5-point scale (1 = never, 5 = always)
Change in Parenting | Baseline; 3 months
  The Alabama Parenting Questionnaire
Intentions to use the PYCC parent training website | Baseline
  1 items taping into parents intentions to use the PYCC parent training website

CONTACTS AND LOCATIONS:
Locations (1):
- Merrill Palmer Skillman Institute, Detroit, Michigan, United States